CLINICAL TRIAL: NCT00314886
Title: Effect of an Enriched Butyrogenic Fibres Diet on Rectal Sensitivity in Healthy Control and IBS Patients.
Brief Title: Effect of Butyrogenic Fibers in IBS Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other); EA 3848 UdA (Unknown); ERT: Clinical Trial Technology Solutions (Other)
Responsible Party: Pr Michel Dapoigny, CHU Clermont-Ferrand
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU63-0009
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Diet; Fiber; Irritable Bowel Syndrome; Colonic Flora
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Diet

SUMMARY:
Despite there being no clearcut advantages, one of the most common recommendations in IBS management is to increase the amount of dietary fibres. In some IBS patients fibres have a deleterious effect on pain and bloating. It has been shown that butyrate can increase colonic sensitivity in rats. Our purpose is to study whether butyrogenic fibres can modify rectal sensitivity and symptoms in IBS and healthy control through a modification of colonic flora.

DETAILED DESCRIPTION:
Despite there being no clearcut advantages, one of the most common recommendations in IBS management is to increase the amount of dietary fibres. In some IBS patients fibres have a deleterious effect on pain and bloating. It has been shown that butyrate can increase colonic sensitivity in rats. Our purpose is to study whether butyrogenic fibres can modify rectal sensitivity and symptoms in IBS and healthy control through a modification of colonic flora.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-60 years
* Normal volunteers and patients with IBS assessed by Rome II criteria
* Effective contraception
* Affiliated to National Health Service
* Having received oral and written information about the study
* Having provided her written informed consent

Exclusion Criteria:

* Significant clinical or biological abnormality
* Organic gastrointestinal disease
* Subjects having lower than 15g/day or higher than 20g/day fibres intake
* Antibiotic treatment during the month preceding the pre inclusion day
* Antispasmodics, antidiarrheics, laxatives, and prokinetics during the week preceding the pre inclusion day and during all the study period.
* Digestive surgery tract except appendectomy and cholecystectomy
* Alcohol abuse
* Drug addiction
* Major psychiatric disorder

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-01; Study Completion 2005-07 (Estimated)

PRIMARY OUTCOMES:
Discomfort threshold to rectal distension

SECONDARY OUTCOMES:
Rectal sensitivity : first sensation and threshold for first sensation of the need to defecate.
Intestinal discomfort (questionnaire)
Quality of life (questionnaire)
Taxonomic composition of colonic flora
Functional composition of colonic flora
Fermentation profile of ingested fibre

CONTACTS AND LOCATIONS:
Overall Officials: Michel Dapoigny, Pr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, Auvergne, France

REFERENCES:
- [Background] Dunlop SP, Spiller RC. Nutritional issues in irritable bowel syndrome. Curr Opin Clin Nutr Metab Care. 2001 Nov;4(6):537-40. doi: 10.1097/00075197-200111000-00013. PMID 11706290
- [Background] Francis CY, Whorwell PJ. Bran and irritable bowel syndrome: time for reappraisal. Lancet. 1994 Jul 2;344(8914):39-40. doi: 10.1016/s0140-6736(94)91055-3. PMID 7912305
- [Background] Harmsen HJ, Raangs GC, He T, Degener JE, Welling GW. Extensive set of 16S rRNA-based probes for detection of bacteria in human feces. Appl Environ Microbiol. 2002 Jun;68(6):2982-90. doi: 10.1128/AEM.68.6.2982-2990.2002. PMID 12039758
- [Background] Jones R, Lydeard S. Irritable bowel syndrome in the general population. BMJ. 1992 Jan 11;304(6819):87-90. doi: 10.1136/bmj.304.6819.87. PMID 1737146
- [Background] Jones VA, McLaughlan P, Shorthouse M, Workman E, Hunter JO. Food intolerance: a major factor in the pathogenesis of irritable bowel syndrome. Lancet. 1982 Nov 20;2(8308):1115-7. doi: 10.1016/s0140-6736(82)92782-9. PMID 6128447
- [Background] King TS, Elia M, Hunter JO. Abnormal colonic fermentation in irritable bowel syndrome. Lancet. 1998 Oct 10;352(9135):1187-9. doi: 10.1016/s0140-6736(98)02146-1. PMID 9777836
- [Background] Snook J, Shepherd HA. Bran supplementation in the treatment of irritable bowel syndrome. Aliment Pharmacol Ther. 1994 Oct;8(5):511-4. doi: 10.1111/j.1365-2036.1994.tb00323.x. PMID 7865643
- [Background] Tarrerias AL, Millecamps M, Alloui A, Beaughard C, Kemeny JL, Bourdu S, Bommelaer G, Eschalier A, Dapoigny M, Ardid D. Short-chain fatty acid enemas fail to decrease colonic hypersensitivity and inflammation in TNBS-induced colonic inflammation in rats. Pain. 2002 Nov;100(1-2):91-7. doi: 10.1016/s0304-3959(02)00234-8. PMID 12435462
- [Background] Bourdu S, Dapoigny M, Chapuy E, Artigue F, Vasson MP, Dechelotte P, Bommelaer G, Eschalier A, Ardid D. Rectal instillation of butyrate provides a novel clinically relevant model of noninflammatory colonic hypersensitivity in rats. Gastroenterology. 2005 Jun;128(7):1996-2008. doi: 10.1053/j.gastro.2005.03.082. PMID 15940632